

## **Informed Consent Form (ICF)**

Validation Study of VIRADIA: A Virtual Reality Diagnostic Platform for the Assessment of Neurological and Cognitive Functions

Protocol ID: 09105-03-804 NCT Number: -Document Date: December 03, 2025

**Sponsor:** Gametherapy s.r.o.

Study Site: INNER s.r.o., Fatranská 873/12, 94901 Nitra, Slovakia

Consent to the processing of personal data under Article 6(1)(a) of Regulation (EU) 2016/679 (GDPR).

I hereby confirm that I have been informed about the purpose, procedures, and nature of the VIRADIA research project, aimed at developing and testing a virtual reality (VR) diagnostic tool for assessing cognitive and motor functions.

The research is conducted by GAMETHERAPY s.r.o., Radlinského 11, 949 01 Nitra, Company ID: 54827655, which is the Data Controller under the GDPR. Personal data will be processed exclusively for research purposes.

I voluntarily consent to the processing of my personal data for the purposes of this research. The following categories of data may be collected:

- 1. Basic personal data such as demographics (age, sex, education, employment) Agree / Do not agree
- 2. Performance data from VR testing (reaction times, movement accuracy) Agree / Do not agree
- 3. Health-related data voluntarily provided by me (neurological conditions) Agree / Do not agree

All data will be pseudonymised using a unique participant ID. Only authorized research staff can link this ID to my identity. Data will not be shared with third parties except authorized persons or contracted processors under Article 28 GDPR.

This consent is valid for the duration of the research project and no longer than 10 years. Data will not be transferred outside the EU.

I acknowledge that the processing follows GDPR and Slovak Act No. 18/2018 Coll. I have been informed of my rights under Articles 12–23 GDPR.

To exercise these rights, I may contact the controller at: viradia@gametherapy.eu

| have read |
|-----------|

| In Nitra, on |
|--------------------------|
| Participant's full name: |
| Signature: |

## Rights of the Data Subject

- Right to withdraw consent You may withdraw consent at any time.
- Right of access You may obtain a copy of your personal data and information about its processing.
- Right to rectification You may request corrections to inaccurate or incomplete data.
- Right to erasure You may request deletion of personal data that is no longer necessary.
- Right to restriction of processing Applies in certain cases.
- Right to data portability You may request transfer of your data to another controller.
- Right to object You may object to processing based on legitimate interests.
- Right to lodge a complaint Office for Personal Data Protection of the Slovak Republic, Námestie 1. mája 7286/18, 811 06 Bratislava; tel.: +421 2 3231 3214; email: statny.dozor@pdp.gov.sk